CLINICAL TRIAL: NCT06484465
Title: Urdu Translation and Psychometric Analysis of Bimanual Functional Classification System BFMF2
Brief Title: Urdu Translation of Bimanaual Fine Motor Functional Classification System 2
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR & AHS/23/0780
Record Dates: First submitted 2024-06-11; First posted 2024-07-03 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Bimanual fine motor classification-2; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2002, Beckung and Hagberg introduced the Bimanual Fine Motor Function (BFMF) classification system. However, the initial version struggled to clearly distinguish between its five defined levels. Despite this, the BFMF system aimed to align with the Gross Motor Function Classification System (GMFCS) levels. Since its introduction, the BFMF system has been widely utilized in the Surveillance of Cerebral Palsy in Europe (SCPE) registry and various epidemiological studies

DETAILED DESCRIPTION:
Beckung and Hagberg developed the Bimanual Fine Motor Function (BFMF) classification system in 2002. Although the initial version had limitations in clearly differentiating between its five levels, it aimed to align with the Gross Motor Function Classification System (GMFCS). Since then, the BFMF system has been widely used in the Surveillance of Cerebral Palsy in Europe (SCPE) registry and various epidemiological studies. The BFMF is a five-level ordinal scale, ranging from Level I (best performance) to Level V (most limited function), designed to assess the ability of children with cerebral palsy to use both hands together to handle objects. Evaluation is based on observation of bimanual performance and parental reports of usual performance. This study consists of two parts: a pilot study for physiotherapists, with defined inclusion and exclusion criteria, and a main study involving cerebral palsy patients, using a finalized Urdu version of the questionnaire to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-15 years
* Gender: Both male and female patients
* Type of CP: Diplegic, athetoid, ataxic, and spastic forms
* Gross Motor Function Classification System (GMFCS) level: 2 or 3

Exclusion Criteria:

* - Orthopedic conditions such as fractures or rickets
* Systemic disorders, including inflammatory diseases and autoimmune conditions
* Psychological and behavioral issues.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: the study focuses on school-aged children with various types of Cerebral Palsy, with moderate to severe gross motor impairments, as classified by the GMFCS system. The study does not include children who have musculoskeletal problems, chronic health conditions, or mental health concerns that may impact their ability to participate or affect the study's outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Bimanual fine motor classification system 2 | 6 months
  Urdu version of Bimanual fine motor classification system 2 The Bimanual Fine Motor Function (BFMF) classifies fine motor function in children with cerebral palsy. The five levels in BFMF form an ordinal scale, which means that the levels are 'ordered' but differences between levels are not necessarily equal, and each level includes children with relatively varied function. It is therefore unlikely that BFMF is sensitive to changes after an intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Samar Mughal, MS*, Principal Investigator — Riphah International University; Tehreem Mukhtar, PhD *, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seyhan-Biyik K, Delioglu K, Tuncdemir M, Unes S, Ozal C, Kerem-Gunel M. Asymmetric involvement of hands: Psychometric properties of the Turkish version of the Bimanual Fine Motor Function 2.0 classification in children with cerebral palsy. J Hand Ther. 2024 Jul-Sep;37(3):429-437. doi: 10.1016/j.jht.2023.08.006. Epub 2023 Sep 28. PMID 37777439